CLINICAL TRIAL: NCT07172919
Title: A Rollover Study of Sotorasib With or Without Panitumumab for the Treatment of Cancer Subjects With KRAS p.G12C Mutation Previously Treated in an Amgen-Sponsored Study
Brief Title: A Rollover Study Evaluating Sotorasib With or Without Panitumumab in Participants With KRAS p.G12C Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250089; 2025-522355-26 (Other: EU CT Number); U1111-1322-4422 (Other: WHO/UTN Number)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; Sotorasib; Panitumumab; AMG 510
MeSH Terms: interventions — sotorasib; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Sotorasib (Experimental): Sotorasib will be administered once daily, orally in 28-day treatment cycles for up to approximately 18 months or until withdrawal of consent, lost to follow-up, or death, whichever occurs first.
  Interventions: Drug: Sotorasib
- Arm B: Sotorasib in Combination with Panitumumab (Experimental): Sotorasib will be administered once daily, orally, in combination with Panitumumab intravenous (IV) infusion every two weeks on Day 1 and Day 15 in 28-day treatment cycles. Treatment will continue for up to approximately 18 months or until withdrawal of consent, lost to follow-up, or death, whichever occurs first.
  Interventions: Drug: Sotorasib; Drug: Panitumumab

INTERVENTIONS:
Drug: Sotorasib — Sotorasib will be administered orally as a tablet.
  Other Names: AMG 510
Drug: Panitumumab — Panitumumab will be administered as an IV infusion.
  Arms: Arm B: Sotorasib in Combination with Panitumumab

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of the continuation of sotorasib with or without panitumumab and/or other anti-cancer therapies in participants continuing to derive benefit in Amgen-sponsored protocols.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥ 18 years.
* Life expectancy of > 3 months, in the opinion of the investigator.
* Ability to take oral medications and willing to record daily adherence to sotorasib through the use of a written diary.
* Participant is currently receiving treatment with sotorasib alone or in combination therapy in an Amgen-sponsored trial that has met its endpoints or otherwise will be stopping (also referred to as parent study) and are continuing to receive clinical benefit in the opinion of the investigator.
* For a participant on combination therapy in their parent study, treatment with other anti-cancer therapies is allowed provided it matches the parent study.
* Eastern Cooperative Oncology Group Performance Status of ≤ 2.

Exclusion Criteria:

* Participant had permanently discontinued from sotorasib study treatment in the parent study before the parent study's completion.
* Ongoing, unresolved toxicity requiring interruption of sotorasib treatment at the time of the termination of the parent study.
* Local access to commercially available investigational product(s) at no cost to the participant as permitted by local/country regulation.
* Anticipated toxicities of sotorasib study treatment outweigh the clinical benefit to the participant in the opinion of the investigator.
* Participant unlikely to be able to complete all protocol-required procedures, restrictions and requirements, in the judgment of the individual and investigator.
* Significant uncontrolled concomitant disease that could affect compliance with protocol procedures or interpretation of results or that pose a risk to participant safety, in the opinion of the investigator.
* Female participants of childbearing potential unwilling to use protocol-specified method of contraception during treatment and for an additional:

  * 7 days after the last dose of sotorasib.
  * 2 months after the last dose of panitumumab.
* Female participants who are breastfeeding or who plan to breastfeed while on study through:

  * 7 days after the last dose of sotorasib.
  * 2 months after the last dose of panitumumab.
* Female participants planning to become pregnant while on study through:

  * 7 days after the last dose of sotorasib.
  * 2 months after the last dose of panitumumab.
* Female participants of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a highly sensitive urine or serum pregnancy test.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 7 days after the last dose of sotorasib.
* Male participants with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 7 days after the last dose of sotorasib.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 7 days after the last dose of sotorasib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 18 months
  Incidence and severity of TEAEs, clinically significant changes in vital signs, and clinical laboratory tests will be reported as TEAEs.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com